CLINICAL TRIAL: NCT01186289
Title: Statin Therapy To Limit Cognitive Dysfunction After Cardiac Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator decided not to pursue enrollment due to changes in standard of care.
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Mark Newman, M. D., Duke University Medical Center Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO00020165
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2011-02

CONDITIONS: Neurocognitive Dysfunction
Keywords: Neurocognitive Dysfunction
MeSH Terms: conditions — Cognition Disorders | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atorvastatin (Experimental): high dose atorvastatin therapy (80 mg/day) beginning 48 to 72-hours preoperatively and continuing until 6-weeks postoperatively
  Interventions: Drug: atorvastatin
- placebo (Placebo Comparator)
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — high dose atorvastatin therapy (80 mg/day) beginning 48 to 72-hours preoperatively and continuing until 6-weeks postoperatively
  Other Names: Lipitor

SUMMARY:
The primary aim of our prospective, randomized, double-blind interventional clinical trial is to determine the effectiveness of high dose atorvastatin therapy to reduce post operative cognitive dysfunction (POCD) in patients undergoing cardiac valve surgery. We hypothesize that therapy with high dose atorvastatin will significantly reduce the incidence and/or severity of POCD.

ELIGIBILITY:
Inclusion Criteria:

* Fifty informed and consenting patients for cardiac valve surgery with CPB , greater than 50 years of age and under the care of one or more of the investigators or consultants will be prospectively enrolled over a one-year period (plus one-year for follow-up).

Exclusion Criteria:

* Patients with a history of the following disease entities will be excluded:

  * symptomatic cerebrovascular disease with substantial residual deficit, alcohol abuse, psychiatric illness, renal failure (creatinine>2.0),
  * hepatic dysfunction (ALT or AST > 1.5 x ULN), history of allergy or myopathy with statin therapy, pregnant or breastfeeding women or other comorbidities that in the opinion of the investigator could limit patient participation. Exclusion criteria are designed to limit confounding and enhance differentiation of deficits related to surgery and or treatment.
  * Patients who are unable to read and thus unable to complete the neurocognitive testing will also be excluded.
  * Patients having concomitant carotid endarterectomy or other vascular surgery will also be excluded to provide a more homogeneous sample for comparison.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Dysfunction | 6 weeks and 1 year post surgery
  The subject will under go a battery of neurological test at baseline, 6 weeks post surgery and at 1 year post surgery to assess neurocognitive status.

CONTACTS AND LOCATIONS:
Overall Officials: Mark F Newman, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Small BJ, Gagnon E, Robinson B. Early identification of cognitive deficits: preclinical Alzheimer's disease and mild cognitive impairment. Geriatrics. 2007 Apr;62(4):19-23. PMID 17408315
- [Background] Small N. Living well until you die: quality of care and quality of life in palliative and dementia care. Ann N Y Acad Sci. 2007 Oct;1114:194-203. doi: 10.1196/annals.1396.019. Epub 2007 Oct 12. PMID 17934058
- [Background] Newman S, Stygall J, Hirani S, Shaefi S, Maze M. Postoperative cognitive dysfunction after noncardiac surgery: a systematic review. Anesthesiology. 2007 Mar;106(3):572-90. doi: 10.1097/00000542-200703000-00023. PMID 17325517
- [Background] Newman MF, Mathew JP, Grocott HP, Mackensen GB, Monk T, Welsh-Bohmer KA, Blumenthal JA, Laskowitz DT, Mark DB. Central nervous system injury associated with cardiac surgery. Lancet. 2006 Aug 19;368(9536):694-703. doi: 10.1016/S0140-6736(06)69254-4. PMID 16920475
- [Background] Tuman KJ, McCarthy RJ, Najafi H, Ivankovich AD. Differential effects of advanced age on neurologic and cardiac risks of coronary artery operations. J Thorac Cardiovasc Surg. 1992 Dec;104(6):1510-7. PMID 1453714
- [Background] Weintraub WS, Jones EL, Craver J, Guyton R, Cohen C. Determinants of prolonged length of hospital stay after coronary bypass surgery. Circulation. 1989 Aug;80(2):276-84. doi: 10.1161/01.cir.80.2.276. PMID 2787709
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Barber PA, Hach S, Tippett LJ, Ross L, Merry AF, Milsom P. Cerebral ischemic lesions on diffusion-weighted imaging are associated with neurocognitive decline after cardiac surgery. Stroke. 2008 May;39(5):1427-33. doi: 10.1161/STROKEAHA.107.502989. Epub 2008 Mar 6. PMID 18323490
- [Background] Cimino M, Gelosa P, Gianella A, Nobili E, Tremoli E, Sironi L. Statins: multiple mechanisms of action in the ischemic brain. Neuroscientist. 2007 Jun;13(3):208-13. doi: 10.1177/1073858406297121. PMID 17519364
- [Background] Rikitake Y, Liao JK. Rho GTPases, statins, and nitric oxide. Circ Res. 2005 Dec 9;97(12):1232-5. doi: 10.1161/01.RES.0000196564.18314.23. PMID 16339495
- [Background] Huang PL, Huang Z, Mashimo H, Bloch KD, Moskowitz MA, Bevan JA, Fishman MC. Hypertension in mice lacking the gene for endothelial nitric oxide synthase. Nature. 1995 Sep 21;377(6546):239-42. doi: 10.1038/377239a0. PMID 7545787
- [Background] Huang Z, Huang PL, Ma J, Meng W, Ayata C, Fishman MC, Moskowitz MA. Enlarged infarcts in endothelial nitric oxide synthase knockout mice are attenuated by nitro-L-arginine. J Cereb Blood Flow Metab. 1996 Sep;16(5):981-7. doi: 10.1097/00004647-199609000-00023. PMID 8784243
- [Background] Huang Z, Huang PL, Panahian N, Dalkara T, Fishman MC, Moskowitz MA. Effects of cerebral ischemia in mice deficient in neuronal nitric oxide synthase. Science. 1994 Sep 23;265(5180):1883-5. doi: 10.1126/science.7522345.
- [Background] Dalkara T, Morikawa E, Panahian N, Moskowitz MA. Blood flow-dependent functional recovery in a rat model of focal cerebral ischemia. Am J Physiol. 1994 Aug;267(2 Pt 2):H678-83. doi: 10.1152/ajpheart.1994.267.2.H678. PMID 8067423
- [Background] Zhang F, Iadecola C. Reduction of focal cerebral ischemic damage by delayed treatment with nitric oxide donors. J Cereb Blood Flow Metab. 1994 Jul;14(4):574-80. doi: 10.1038/jcbfm.1994.71. PMID 8014203
- [Background] Morikawa E, Huang Z, Moskowitz MA. L-arginine decreases infarct size caused by middle cerebral arterial occlusion in SHR. Am J Physiol. 1992 Nov;263(5 Pt 2):H1632-5. doi: 10.1152/ajpheart.1992.263.5.H1632. PMID 1443214
- [Background] Endres M, Laufs U, Huang Z, Nakamura T, Huang P, Moskowitz MA, Liao JK. Stroke protection by 3-hydroxy-3-methylglutaryl (HMG)-CoA reductase inhibitors mediated by endothelial nitric oxide synthase. Proc Natl Acad Sci U S A. 1998 Jul 21;95(15):8880-5. doi: 10.1073/pnas.95.15.8880. PMID 9671773
- [Background] Carloni S, Mazzoni E, Cimino M, De Simoni MG, Perego C, Scopa C, Balduini W. Simvastatin reduces caspase-3 activation and inflammatory markers induced by hypoxia-ischemia in the newborn rat. Neurobiol Dis. 2006 Jan;21(1):119-26. doi: 10.1016/j.nbd.2005.06.014. Epub 2005 Jul 27. PMID 16054375
- [Background] Sironi L, Banfi C, Brioschi M, Gelosa P, Guerrini U, Nobili E, Gianella A, Paoletti R, Tremoli E, Cimino M. Activation of NF-kB and ERK1/2 after permanent focal ischemia is abolished by simvastatin treatment. Neurobiol Dis. 2006 May;22(2):445-51. doi: 10.1016/j.nbd.2005.12.004. Epub 2006 Feb 9. PMID 16480888
- [Background] Weber C, Erl W, Weber KS, Weber PC. HMG-CoA reductase inhibitors decrease CD11b expression and CD11b-dependent adhesion of monocytes to endothelium and reduce increased adhesiveness of monocytes isolated from patients with hypercholesterolemia. J Am Coll Cardiol. 1997 Nov 1;30(5):1212-7. doi: 10.1016/s0735-1097(97)00324-0. PMID 9350917
- [Background] Elkind MS. Inflammation, atherosclerosis, and stroke. Neurologist. 2006 May;12(3):140-8. doi: 10.1097/01.nrl.0000215789.70804.b0. PMID 16688015
- [Background] Freedman JE, Loscalzo J, Barnard MR, Alpert C, Keaney JF, Michelson AD. Nitric oxide released from activated platelets inhibits platelet recruitment. J Clin Invest. 1997 Jul 15;100(2):350-6. doi: 10.1172/JCI119540. PMID 9218511
- [Background] Laufs U, Gertz K, Huang P, Nickenig G, Bohm M, Dirnagl U, Endres M. Atorvastatin upregulates type III nitric oxide synthase in thrombocytes, decreases platelet activation, and protects from cerebral ischemia in normocholesterolemic mice. Stroke. 2000 Oct;31(10):2442-9. doi: 10.1161/01.str.31.10.2442. PMID 11022078
- [Background] Labios M, Martinez M, Gabriel F, Guiral V, Martinez E, Aznar J. Effect of atorvastatin upon platelet activation in hypercholesterolemia, evaluated by flow cytometry. Thromb Res. 2005;115(4):263-70. doi: 10.1016/j.thromres.2004.08.016. PMID 15668185
- [Background] Hwang YS, Tsai WC, Lu YH, Lin CC, Chen YF. Effect of atorvastatin on the expression of CD40 ligand and P-selectin on platelets in patients with hypercholesterolemia. Am J Cardiol. 2004 Aug 1;94(3):364-6. doi: 10.1016/j.amjcard.2004.04.037. PMID 15276107
- [Background] Asahi M, Huang Z, Thomas S, Yoshimura S, Sumii T, Mori T, Qiu J, Amin-Hanjani S, Huang PL, Liao JK, Lo EH, Moskowitz MA. Protective effects of statins involving both eNOS and tPA in focal cerebral ischemia. J Cereb Blood Flow Metab. 2005 Jun;25(6):722-9. doi: 10.1038/sj.jcbfm.9600070. PMID 15716855
- [Background] LaRosa JC, Grundy SM, Waters DD, Shear C, Barter P, Fruchart JC, Gotto AM, Greten H, Kastelein JJ, Shepherd J, Wenger NK; Treating to New Targets (TNT) Investigators. Intensive lipid lowering with atorvastatin in patients with stable coronary disease. N Engl J Med. 2005 Apr 7;352(14):1425-35. doi: 10.1056/NEJMoa050461. Epub 2005 Mar 8. PMID 15755765
- [Background] Waters DD, LaRosa JC, Barter P, Fruchart JC, Gotto AM Jr, Carter R, Breazna A, Kastelein JJ, Grundy SM. Effects of high-dose atorvastatin on cerebrovascular events in patients with stable coronary disease in the TNT (treating to new targets) study. J Am Coll Cardiol. 2006 Nov 7;48(9):1793-9. doi: 10.1016/j.jacc.2006.07.041. Epub 2006 Oct 17. PMID 17084252
- [Background] Muldoon MF, Barger SD, Ryan CM, Flory JD, Lehoczky JP, Matthews KA, Manuck SB. Effects of lovastatin on cognitive function and psychological well-being. Am J Med. 2000 May;108(7):538-46. doi: 10.1016/s0002-9343(00)00353-3. PMID 10806282
- [Background] Harrison RW, Ashton CH. Do cholesterol-lowering agents affect brain activity? A comparison of simvastatin, pravastatin, and placebo in healthy volunteers. Br J Clin Pharmacol. 1994 Mar;37(3):231-6. doi: 10.1111/j.1365-2125.1994.tb04268.x. PMID 8198930
- [Background] Mathew JP, Grocott HP, McCurdy JR, Ti LK, Davis RD, Laskowitz DT, Podgoreanu MV, Swaminathan M, Lynch J, Stafford-Smith M, White WD, Newman MF. Preoperative statin therapy does not reduce cognitive dysfunction after cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2005 Jun;19(3):294-9. doi: 10.1053/j.jvca.2005.03.004. PMID 16130053
- [Background] Parale GP, Baheti NN, Kulkarni PM, Panchal NV. Effects of atorvastatin on higher functions. Eur J Clin Pharmacol. 2006 Apr;62(4):259-65. doi: 10.1007/s00228-005-0073-z. Epub 2006 Feb 18. PMID 16489473
- [Background] LaRosa JC, Grundy SM, Kastelein JJ, Kostis JB, Greten H; Treating to New Targets (TNT) Steering Committee and Investigators. Safety and efficacy of Atorvastatin-induced very low-density lipoprotein cholesterol levels in Patients with coronary heart disease (a post hoc analysis of the treating to new targets [TNT] study). Am J Cardiol. 2007 Sep 1;100(5):747-52. doi: 10.1016/j.amjcard.2007.03.102. Epub 2007 Jun 14. PMID 17719314
- [Background] Schouten O, Boersma E, Hoeks SE, Benner R, van Urk H, van Sambeek MR, Verhagen HJ, Khan NA, Dunkelgrun M, Bax JJ, Poldermans D; Dutch Echocardiographic Cardiac Risk Evaluation Applying Stress Echocardiography Study Group. Fluvastatin and perioperative events in patients undergoing vascular surgery. N Engl J Med. 2009 Sep 3;361(10):980-9. doi: 10.1056/NEJMoa0808207. PMID 19726772
- [Background] Davidson MH, Robinson JG. Safety of aggressive lipid management. J Am Coll Cardiol. 2007 May 1;49(17):1753-62. doi: 10.1016/j.jacc.2007.01.067. Epub 2007 Apr 16. PMID 17466224
- [Background] Mariscalco G, Lorusso R, Klersy C, Ferrarese S, Tozzi M, Vanoli D, Domenico BV, Sala A. Observational study on the beneficial effect of preoperative statins in reducing atrial fibrillation after coronary surgery. Ann Thorac Surg. 2007 Oct;84(4):1158-64. doi: 10.1016/j.athoracsur.2007.05.021. PMID 17888963
- [Background] Coleman CI, Lucek DM, Hammond J, White CM. Preoperative statins and infectious complications following cardiac surgery. Curr Med Res Opin. 2007 Aug;23(8):1783-90. doi: 10.1185/030079907X210570. PMID 17597556
- [Background] Kulik A, Levin R, Ruel M, Mesana TG, Solomon DH, Choudhry NK. Patterns and predictors of statin use after coronary artery bypass graft surgery. J Thorac Cardiovasc Surg. 2007 Oct;134(4):932-8. doi: 10.1016/j.jtcvs.2007.05.039. PMID 17903510
- [Background] Filion KB, Pilote L, Rahme E, Eisenberg MJ. Perioperative use of cardiac medical therapy among patients undergoing coronary artery bypass graft surgery: a systematic review. Am Heart J. 2007 Sep;154(3):407-14. doi: 10.1016/j.ahj.2007.04.036. PMID 17719282
- [Background] Patti G, Pasceri V, Colonna G, Miglionico M, Fischetti D, Sardella G, Montinaro A, Di Sciascio G. Atorvastatin pretreatment improves outcomes in patients with acute coronary syndromes undergoing early percutaneous coronary intervention: results of the ARMYDA-ACS randomized trial. J Am Coll Cardiol. 2007 Mar 27;49(12):1272-8. doi: 10.1016/j.jacc.2007.02.025. PMID 17394957
- [Background] Patti G, Chello M, Pasceri V, Colonna D, Nusca A, Miglionico M, D'Ambrosio A, Covino E, Di Sciascio G. Protection from procedural myocardial injury by atorvastatin is associated with lower levels of adhesion molecules after percutaneous coronary intervention: results from the ARMYDA-CAMs (Atorvastatin for Reduction of MYocardial Damage during Angioplasty-Cell Adhesion Molecules) substudy. J Am Coll Cardiol. 2006 Oct 17;48(8):1560-6. doi: 10.1016/j.jacc.2006.06.061. Epub 2006 Sep 26. PMID 17045888
- [Background] Pasceri V, Patti G, Nusca A, Pristipino C, Richichi G, Di Sciascio G; ARMYDA Investigators. Randomized trial of atorvastatin for reduction of myocardial damage during coronary intervention: results from the ARMYDA (Atorvastatin for Reduction of MYocardial Damage during Angioplasty) study. Circulation. 2004 Aug 10;110(6):674-8. doi: 10.1161/01.CIR.0000137828.06205.87. Epub 2004 Jul 26. PMID 15277322
- [Background] Ruff RM, Parker SB. Gender- and age-specific changes in motor speed and eye-hand coordination in adults: normative values for the Finger Tapping and Grooved Pegboard Tests. Percept Mot Skills. 1993 Jun;76(3 Pt 2):1219-30. doi: 10.2466/pms.1993.76.3c.1219. PMID 8337069
- [Background] Murkin JM, Stump DA, Blumenthal JA, McKhann G. Defining dysfunction: group means versus incidence analysis--a statement of consensus. Ann Thorac Surg. 1997 Sep;64(3):904-5. doi: 10.1016/s0003-4975(97)00743-1. No abstract available. PMID 9307516
- [Background] Murkin JM, Newman SP, Stump DA, Blumenthal JA. Statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery. Ann Thorac Surg. 1995 May;59(5):1289-95. doi: 10.1016/0003-4975(95)00106-u. No abstract available. PMID 7733754
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Newman MF, Croughwell ND, Blumenthal JA, White WD, Lewis JB, Smith LR, Frasco P, Towner EA, Schell RM, Hurwitz BJ, et al. Effect of aging on cerebral autoregulation during cardiopulmonary bypass. Association with postoperative cognitive dysfunction. Circulation. 1994 Nov;90(5 Pt 2):II243-9. PMID 7955260
- [Background] Pahan K, Sheikh FG, Namboodiri AM, Singh I. Lovastatin and phenylacetate inhibit the induction of nitric oxide synthase and cytokines in rat primary astrocytes, microglia, and macrophages. J Clin Invest. 1997 Dec 1;100(11):2671-9. doi: 10.1172/JCI119812. PMID 9389730
- [Background] Rey A. L'examen clinique en psychologie. Paris: Presses Universitaires de France;1964
- [Background] Wechsler D. The Wechsler Adult Intelligence Scale-Revised (WAIS-R). San Antonio, Texas: The Psychological Corporation; 1981
- [Background] Reitan RM. Validity of the trail making test as an indicator of organic brain damage. Percept Mot Skills. 1958;8:271-276.
- [Background] Benton AL, Hansher K. Multilingual Aphasia Examination. Iowa City: University of Iowa Press; 1978
- [Background] Hlatky MA, Bacon C, Boothroyd D, Mahanna E, Reves JG, Newman MF, Johnstone I, Winston C, Brooks MM, Rosen AD, Mark DB, Pitt B, Rogers W, Ryan T, Wiens R, Blumenthal JA. Cognitive function 5 years after randomization to coronary angioplasty or coronary artery bypass graft surgery. Circulation. 1997 Nov 4;96(9 Suppl):II-11-4; discussion II-15. PMID 9386068
- [Background] Fillenbaum GG. Multidimensional functional assessment of older adults (The Duke Older Americans Resources and Services Procedures). Hillsdale, N.J.: Erlbaum Associates; 1988
- [Background] Ware JE, Snow KK, Kosinski M, et al. SF-36 Health Survey: Manual and Interpretation Guide. Lincon, Rhode Island: Qualitymetric, Inc.;2000
- [Background] Ware JE, Kosinski KK, Keller SD. SF-36 Physical and Mental Health Summary Scales: A User's Manual. Boston: Health Assessment Lab, New England Medical Center; 1994
- [Background] Axelrad KJ. Locus of Control and Casual Attributions As they Relate to Expectations for Coping With A Heart Attack. Los Angeles, California School of Professional Psychology; 1981.
- [Background] Radloff LS. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psycological Measures. Vol 1; 1977:385-401.
- [Background] Spielberger C, Gorsuch R, Lushene R. STAI Manual Palo Alto: Consulting Psychologists Press, Inc; 1970
- [Background] Blumenthal JA, Burg MM, Barefoot J, Williams RB, Haney T, Zimet G. Social support, type A behavior, and coronary artery disease. Psychosom Med. 1987 Jul-Aug;49(4):331-40. doi: 10.1097/00006842-198707000-00002. PMID 3615762
- [Background] McNair DM, Kahn RJ. Self-assessment of Cognitive Deficits. In: Crook T., Ferris, S.,Bartus, R., ed. Assessment In Geriatric Psychopharmacology. New Canaan, Ct.: Mark Powley Associates, Inc.: 1983.
- [Background] Rosengarten B, Auch D, Kaps M. Effects of initiation and acute withdrawal of statins on the neurovascular coupling mechanism in healthy, normocholesterolemic humans. Stroke. 2007 Dec;38(12):3193-7. doi: 10.1161/STROKEAHA.107.491423. Epub 2007 Oct 25. PMID 17962596
- [Background] Blanco M, Nombela F, Castellanos M, Rodriguez-Yanez M, Garcia-Gil M, Leira R, Lizasoain I, Serena J, Vivancos J, Moro MA, Davalos A, Castillo J. Statin treatment withdrawal in ischemic stroke: a controlled randomized study. Neurology. 2007 Aug 28;69(9):904-10. doi: 10.1212/01.wnl.0000269789.09277.47. PMID 17724294
- [Background] Cronbach LJ. Essentials of Psychological Testing. New York: Harper and Row; 1970